CLINICAL TRIAL: NCT04027816
Title: Protocol RT001-009: A Natural History Study of Infantile Neuroaxonal Dystrophy
Brief Title: A Natural History Study of Infantile Neuroaxonal Dystrophy
Status: Completed | Type: Observational
Sponsor: Biojiva LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: RT001-009
Record Dates: First submitted 2019-07-16; First posted 2019-07-22 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Neuroaxonal Dystrophy, Infantile
Keywords: PLA2G6-related NBIA; INAD; PLA2G6
MeSH Terms: conditions — Neuroaxonal Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a longitudinal and prospective study of the natural history of infantile neuroaxonal dystrophy (INAD).

DETAILED DESCRIPTION:
After obtaining informed consent, the study participants' relevant medical records will be collected and reviewed for this study. Next, a clinic visit will be scheduled with the patient's family and an observing MD/DO/MBBS from a sponsor site to confirm and clarify information in the medical records.

A baseline evaluation of clinical status will also be performed during this visit to serve as visit one in this longitudinal, prospective natural history study. Subsequent visits will take place every 6 months, for up to 24 months. Key components of this prospective study at each visit include a neurodevelopment exam tailored for INAD, application of the CHOP-INTEND neurodevelopment scale, the Hammersmith infant neurological examination and the modified Ashworth spasticity scale as well as collection of monthly parental severity scoring and monthly home videos of activities of daily living (ADLs).

Data from this study will be pooled and presented in aggregate, without identification of individual subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 months to 10 years of age
* Medical history consistent with the symptoms of classic INAD (onset of symptoms between the ages of 6 months and 3 years)
* Homozygous or compound heterozygous PLA2G6 variants
* Signed informed consent form (ICF) prior to entry into the registry

Exclusion Criteria:

* Diagnosis of atypical NAD (ANAD)
* Additional underlying diagnosis with features that overlap with INAD
* Unwilling or unable to allow medical record review
* Unwilling or unable to participate in serial assessments every 6 months (including deceased patients)

Ages: 18 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Living males or females with a diagnosis of classic INAD between 18 months to 10 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
INAD Mortality | 1-2 years of follow-up is planned
  Overall analysis

SECONDARY OUTCOMES:
INAD Morbidity | 1-2 years of follow-up is planned
  Videotaped, structured neurological assessment
INAD Morbidity | 1-2 years of follow-up is planned
  CHOP-INTEND Neuro-development Score
INAD Morbidity | 1-2 years of follow-up is planned
  Hammersmith infant neurological examination
INAD morbidity | 1-2 years of follow-up is planned
  Modified Ashworth spasticity scale

CONTACTS AND LOCATIONS:
Overall Officials: Peter Milner, MD, Study Director — Biojiva LLC
Locations (5):
- Peking University First Hospital, Beijing, China
- National Research Centre, Cairo, Egypt
- EN1 Neuro Services Pvt. Ltd, Mumbai, India
- King Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia
- National Institute of Neurology of Tunis, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No